CLINICAL TRIAL: NCT04089059
Title: A Prospective, Multi-Center, Open Label, Single Arm Clinical Trial Evaluating the Safety and Efficacy of the Cordella™ Pulmonary Artery Sensor System in NYHA Class III Heart Failure Patients (PROACTIVE- HF Trial)
Brief Title: PROACTIVE-HF IDE Trial Heart Failure NYHA Class III
Acronym: PROACTIVE-HF
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Endotronix, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: ETX-HFS-PA-03
Record Dates: First submitted 2019-08-30; First posted 2019-09-13 (Actual); Results first posted 2025-03-03 (Actual); Last update posted 2025-03-03 (Actual); Status verified 2024-12

CONDITIONS: Heart Failure NYHA Class III
Keywords: Heart Failure; Heart Disease; Cardiovascular Disease; Pulmonary Artery Pressure
MeSH Terms: conditions — Heart Failure; Heart Diseases; Cardiovascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Treatment Arm (Other): Pulmonary Artery Pressure Guided Heart Failure Management (PAPGHFM) and Guideline Directed Medical Therapy (GDMT) considering daily Pulmonary Artery Pressure (PAP) measurements and vital signs collected by Cordella Heart Failure System (CHFS).
  Interventions: Device: Cordella™ Pulmonary Artery Sensor System

INTERVENTIONS:
Device: Cordella™ Pulmonary Artery Sensor System — The Cordella PA Sensor System (CorPASS) is intended to measure, record, and transmit pulmonary artery pressure (PAP) data from NYHA Class III heart failure patients at home to clinicians for assessment and patient-centered heart failure management and comprises of seven subsystems that operate together to take daily Pulmonary Artery Pressure (PAP) readings at a patient's home and transmit the results to a care provider for evaluation.
  1. Cordella Sensor
  2. Cordella Delivery System
  3. myCordella Patient Reader
  4. Reader Dock
  5. Cordella Calibration Equipment (CalEQ)
  6. myCordella Hub
  7. Cordella Data Analysis Platform (CDAP)

SUMMARY:
This is a prospective, open- label, single arm, multicenter clinical trial to evaluate the safety and effectiveness of the Cordella PA Sensor System in NYHA Class III Heart Failure Patients compared to a Performance Goal (PG).

ELIGIBILITY:
Inclusion Criteria

1. Subject has given written informed consent
2. Male or female, at least 18 years of age
3. Diagnosis and treatment of HF (regardless of left ventricular ejection fraction (LVEF)) for ≥ 3 months and NYHA Class III HF at time of Screening
4. Subjects should be on stable, optimally titrated medical therapy for at least 30 days, as recommended according to current American Heart Association (AHA)/American College of Cardiology (ACC) guidelines as standard-of-care for HF therapy in the United States, or current European Society of Cardiology (ESC) guidelines for HF treatment in Europe, with any intolerance documented.
5. HF related hospitalization, HF treatment in a hospital day-care setting, or urgent outpatient clinic HF visit for IV diuretics within 12 month (last hospitalization should be 30 days before Screening/Enrollment) and/or N-terminal pro B-type Natriuretic Peptide (NT proBNP) at time of Screening/ Enrollment defined as:

   1. Subjects with LVEF ≤ 50%: NT-proBNP ≥ 1500 pg/mL.
   2. Subjects with LVEF > 50%: NT-proBNP ≥ 800 pg/mL . Thresholds for NT-proBNP (for both LVEF ≤ 50% and LVEF > 50%) will be corrected for body mass index (BMI) using a 4% reduction per BMI unit over 25 kg/m2
6. Subjects should be on diuretic therapy
7. Subjects who are physically able to hold the myCordella™ Patient Reader unit (approximate weight 1.3lb) against the ventral thoracic surface for up to 2 minutes per day while in a seated position, as well as dock and undock the myCordella™ Patient Reader
8. Subjects with sufficient eyesight, hearing, and mental capacity to respond to the myCordella™ Patient Reader's audio/visual cues and operate the myCordella™ Patient Reader
9. Subject has sufficient Cellular and/ or Wi- Fi Internet coverage at home
10. Subject agrees to return to the treating Investigator for all scheduled follow up visits and can return to the hospital for follow up

Exclusion Criteria

1. Intolerance to all neuro-hormonal antagonists (i.e., intolerance to ACE-I, ARB, ARNI, and beta-blockers) due to hypotension or renal dysfunction
2. ACC/AHA Stage D refractory HF (including having received or currently receiving pharmacologic circulatory support with inotropes)
3. Subjects with history of recurrent pulmonary embolism ( ≥2 episodes within 5 years prior to Screening Visit) and/or deep vein thrombosis (< 3 month prior to Screening Visit)
4. Subjects who have had a major cardiovascular (CV) event (e.g. myocardial infarction, stroke) within 3 months of the Screening Visit
5. Unrepaired severe valvular disease
6. Subjects with significant congenital heart disease that has not been repaired and would prevent implantation of the Cordella PA sensor or mechanical/tissue right heart valve(s)
7. Subjects with known coagulation disorders
8. Subjects with a hypersensitivity or allergy to platelet aggregation inhibitors including aspirin, clopidogrel, prasugrel, and ticagrelor; or patients unable to take dual antiplatelet or anticoagulants for one-month post implant
9. Known history of life threatening allergy to contrast dye
10. Subjects whereby RHC is contraindicated
11. Subjects with an active infection at the Sensor Implant Visit
12. Subjects with a Glomerular Filtration Rate (GFR) <25 ml/min or who are on chronic renal dialysis
13. Implanted with Cardiac Resynchronization Therapy (CRT)-Pacemaker (CRT-P) or CRT-Defibrillator (CRT-D) for less than 90 days prior to screening visit
14. Received or are likely to receive an advanced therapy (e.g. mechanical circulatory support or lung or heart transplant) in the next 12 months
15. Subjects who are pregnant or breastfeeding
16. Subjects who are unwilling or deemed by the Investigator to be unwilling to comply with the study protocol, or subjects with a history of non-compliance
17. Severe illness, other than heart disease, which would limit survival to <1 year
18. Subjects whose clinical condition, in the opinion of the Investigator, makes them an unsuitable candidate for the study
19. Subjects enrolled in another investigational trial with an active treatment arm
20. Subject who is in custody by order of an authority or a court of law

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 738 (Actual)
Dates: Start 2020-01-10 (Actual); Primary Completion 2028-04 (Estimated); Study Completion 2028-04 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Sauerland, Study Director — Endotronix, Inc.
Locations (74):
- United States (70):
  - Ascension St Vincent's, Birmingham, Alabama
  - Huntsville Hospital, Huntsville, Alabama
  - Phoenix Cardiovascular Research Group/Insight, Phoenix, Arizona
  - Loma Linda University, Loma Linda, California
  - Eisenhower Medical Center, Rancho Mirage, California
  - UCSD, San Diego, California
  - Kaiser San Francisco, San Francisco, California
  - UCSF Medical Center, San Francisco, California
  - Kaiser Santa Clara, Santa Clara, California
  - South Denver Cardiology, Littleton, Colorado
  - Hartford Hospital, Hartford, Connecticut
  - Baptist Health South Florida, Miami, Florida
  - Ascension Sacred Heart, Pensacola, Florida
  - USF Health, Tampa, Florida
  - Cleveland Clinic, Weston, Florida
  - Piedmont Athens, Athens, Georgia
  - Queens Medical Center, Honolulu, Hawaii
  - Northwestern, Chicago, Illinois
  - U of Chicago, Chicago, Illinois
  - Heart Centers of Illinois, Palos Park, Illinois
  - OSF Healthcare, Peoria, Illinois
  - Ascension St Vincent's, Indianapolis, Indiana
  - University of Iowa Medical Center, Iowa City, Iowa
  - University of Kansas Medical Center (KUMC), Kansas City, Kansas
  - University Of Louisville, Louisville, Kentucky
  - Ochsner Medical Center, New Orleans, Louisiana
  - University of Maryland, Baltimore, Maryland
  - Medstar, Baltimore, Maryland
  - Tufts Medical Center, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center (BIDMC), Boston, Massachusetts
  - Brigham and Women's Hospital (Mass General Brigham), Boston, Massachusetts
  - Henry Ford Hospital, Detroit, Michigan
  - Minneapolis Heart Institute Foundation, Minneapolis, Minnesota
  - University of Minnesota, Minneapolis, Minnesota
  - Centra Care Heart Center, Saint Cloud, Minnesota
  - St. Lukes/ Mid-American Heart Institute, Kansas City, Missouri
  - Hackensack University Medical Center, Hackensack, New Jersey
  - The Valley Hospital, Ridgewood, New Jersey
  - Mount Sinai, New York, New York
  - NYU Langone Health, New York, New York
  - New York Presbyterian Queens, Queens, New York
  - Stony Brook University Med Center, Stony Brook, New York
  - University of Cincinnati, Cincinnati, Ohio
  - Ohio State University, Columbus, Ohio
  - Oregon Health Science Portland, Portland, Oregon
  - Thomas Jefferson Abington, Abington, Pennsylvania
  - Penn State Health, Hershey, Pennsylvania
  - Penn Medicine, Philadelphia, Pennsylvania
  - Thomas Jefferson, Philadelphia, Pennsylvania
  - UPMC, Pittsburgh, Pennsylvania
  - PRISMA Midlands - Palmetto, Columbia, South Carolina
  - PRISMA Health- Upstate, Greenville, South Carolina
  - Sanford, Sioux Falls, South Dakota
  - Tennova Healthcare (Turkey Creek Medical Center), Knoxville, Tennessee
  - Vanderbilt, Nashville, Tennessee
  - Austin Heart, Austin, Texas
  - Craig Cardiovascular Center, Gonzales, Texas
  - Baylor/Texas Heart, Houston, Texas
  - Houston Methodist, Houston, Texas
  - University of Texas/Hermann Memorial, Houston, Texas
  - Baylor - Round Rock, Round Rock, Texas
  - Methodist Healthcare System, San Antonio, Texas
  - Baylor - Temple, Temple, Texas
  - University of Vermont, Burlington, Vermont
  - Sentara Healthcare, Norfolk, Virginia
  - Valley Health System/Winchester Medical Center, Winchester, Virginia
  - University of Washington, Seattle, Washington
  - Providence Health Care, Spokane, Washington
  - West Virginia University, Morgantown, West Virginia
  - University of Wisconsin, Madison, Wisconsin
- Belgium (3):
  - Cardiovascular Center OLV Aalst, Aalst
  - ZNA Middlheim, Antwerp
  - Ziekenhuis- Oost Limburg, Genk
- University Hospital Galway, Galway, Ireland

REFERENCES:
- [Derived] Pourafshar N, Daneshmand A, Karimi A, Wilcox CS. Methods for the Assessment of Volume Overload and Congestion in Heart Failure. Kidney360. 2024 Oct 1;5(10):1584-1593. doi: 10.34067/KID.0000000000000553. Epub 2024 Aug 20. PMID 39480670
- [Derived] Guichard JL, Bonno EL, Nassif ME, Khumri TM, Miranda D, Jonsson O, Shah H, Alexy T, Macaluso GP, Sur J, Hickey G, McCann P, Cowger JA, Badiye A, Old WD, Raza Y, Masha L, Kunavarapu CR, Bennett M, Sharif F, Kiernan M, Mullens W, Chaparro SV, Mahr C, Amin RR, Stevenson LW, Hiivala NJ, Owens MM, Sauerland A, Forouzan O, Klein L. Seated Pulmonary Artery Pressure Monitoring in Patients With Heart Failure: Results of the PROACTIVE-HF Trial. JACC Heart Fail. 2024 Nov;12(11):1879-1893. doi: 10.1016/j.jchf.2024.05.017. Epub 2024 Aug 14. PMID 39152983

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment was initiated on January 10, 2020, and completed on March 9, 2023, among 77 sites in the United States and five (5) sites in Ireland and Belgium. The last implant procedure was performed on March 31, 2023. The patient population consisted of male and female patients, ≥ 18 years of age with a diagnosis of NYHA Class III HF who met the study patient selection criteria.
Pre-assignment Details: Of the 738 enrolled subjects, 528 received an implant, 125 had screen failure and 85 were withdrawn prior to implant. Of 85 withdrawn subjects, in 37 instances the implant procedure was aborted prior to deploying the implant. Of 528 subjects implanted, 72 were in the control group (eliminated in trial redesign). The remaining 456 patients form the mITT population, which was used for all efficacy analyses. All safety analyses used the ITT population (456 mITT + 37 withdrawn = 493 patients).
Groups:
- Former Control Arm: Received standard of care heart failure management (i.e., Guideline Directed Medical Therapy) using the Cordella Heart Failure System (CHFS) excluding the PA pressure sensor until the trial redesign. After trial redesign were crossed over to receive standard of care HF management using the Cordella HF system with the PA pressure sensor.
- Former Treatment Arm: Received standard of care HF management using the Cordella Heart Failure System (CHFS) and Pulmonary Artery Pressure Guided Heart Failure Management (PAPGHFM) using the Cordella Heart Failure System (CHFS) with the PA pressure sensor before and after trial redesign.
- Open Label Arm: Recruited after trial redesign. Received standard of care HF management using the Cordella Heart Failure System (CHFS) and Pulmonary Artery Pressure Guided Heart Failure Management (PAPGHFM) using the Cordella Heart Failure System (CHFS) with the PA pressure sensor.
Period: Overall Study
Arm/Group | Former Control Arm | Former Treatment Arm | Open Label Arm
Started | 72 | 88 | 368
Completed | 66 | 82 | 343
Not Completed | 6 | 6 | 25

BASELINE CHARACTERISTICS:
Population: This table reports the baseline information for the Modified Intent-to-Treat (mITT) population, which was made up of the treatment arm prior to the trial redesign and the open label arm, which received treatment after the trial redesign. The mITT population is the primary cohort for all efficacy analyses. Additionally, the control arm from prior to the trial redesign is reported, who were implanted but did not receive treatment using the implant.
Groups:
- Modified Intent-to-Treat (mITT): Received standard of care heart failure management (i.e., Guideline Directed Medical Therapy) and Pulmonary Artery Pressure Guided Heart Failure Management (PAPGHFM) using the Cordella Heart Failure System (CHFS) with the PA pressure sensor. Made up of open label arm plus former treatment arm.
  Cordella™ Pulmonary Artery Sensor System: The Cordella PA Sensor System (CorPASS) is intended to measure, record, and transmit pulmonary artery pressure (PAP) data from NYHA Class III heart failure patients at home to clinicians for assessment and patient-centered heart failure management and comprises of seven subsystems that operate together to take daily Pulmonary Artery Pressure (PAP) readings at a patient's home and transmit the results to a care provider for evaluation.
  1. Cordella Sensor
  2. Cordella Delivery System
  3. myCordella Patient Reader
  4. Reader Dock
  5. Cordella Calibration Equipment (CalEQ)
  6. myCordella Hub
  7. Cordella Data Analysis Platform (CDAP)
- Total: Total of all reporting groups
Arm/Group | Modified Intent-to-Treat (mITT) | Former Control Arm | Total
Number analyzed (Participants) | 456 | 72 | 528
Age, Continuous [Mean (Standard Deviation); unit: Years] | 63.5 (12.53) | 65.9 (11.26) | 63.8 (12.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 180 | 30 | 210
  Male | 276 | 42 | 318
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 20 | 5 | 25
  Not Hispanic or Latino | 401 | 61 | 462
  Unknown or Not Reported | 35 | 6 | 41
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 1 | 3
  Asian | 7 | 0 | 7
  Native Hawaiian or Other Pacific Islander | 3 | 1 | 4
  Black or African American | 84 | 11 | 95
  White | 347 | 56 | 403
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 13 | 3 | 16
Region of Enrollment [Number; unit: participants]
  Belgium | 12 | 0 | 12
  United States | 438 | 72 | 510
  Ireland | 6 | 0 | 6

OUTCOME MEASURES:

1. Primary Outcome: Efficacy 6 Month Incidence of HF Related Hospitalizations (HFH) or All-cause Mortality
Description: The primary efficacy endpoint was the 6-month incidence of HF related hospitalizations or all-cause mortality in the modified Intent-to-Treat (mITT) population. As per the approved protocol/CIP, for study success the upper confidence bound of the observed event rate in the mITT population was required to be less than the performance goal (PG) of 0.43 events per patient 6-month, or equivalently, the corresponding p-value from the hypothesis test of 6-month incidence rate compared to PG was less than 0.025. Furthermore, the observed incidence rate was required to be less than 0.37. The 6-month incidence rate was derived using a Poisson regression with the number of events as the dependent variable and the exposure time as an offset term. In these analyses, a subject's exposure time was defined as the time to death, early study discontinuation, or 6 months (whichever occurred first).
Time Frame: 6 months
Population: The Modified Intent-to-Treat Population (mITT) includes all implanted subjects from the Open Label Arm and Former Treatment Arm. All primary and secondary effectiveness analyses are performed on the mITT.
Measure: Number (95% Confidence Interval); unit: Events Per Patient Per 6 Months
Groups:
- Modified Intent-to-Treat (mITT): Received standard of care heart failure management (i.e., Guideline Directed Medical Therapy) and Pulmonary Artery Pressure Guided Heart Failure Management (PAPGHFM) using the Cordella Heart Failure System (CHFS) with the PA pressure sensor. Made up of open label arm plus former treatment arm.
Arm/Group | Modified Intent-to-Treat (mITT) | Former Control Arm
Number analyzed (Participants) | 456 | 72
Events Per Patient Per 6 Months | 0.1549 [0.1225 to 0.1957] | 0.2787 [0.1798 to 0.4320]
Statistical Analysis 1: Comparison: Modified Intent-to-Treat (mITT); Test type: Superiority — Poisson regression for comparison of incidence rate against performance goal (0.43); p < 0.0001, Poisson Regression

2. Primary Outcome: Safety: Freedom From Device/System Related Complication
Description: A device/system related complication (DSRC) is defined as an AE that is, or is possibly, related to the device/system (Cordella PA Sensor or electronic components) and is either treated invasively (other than intramuscular medication or diagnostic RHC) or results in subject´s death or explant of the device. The first primary safety endpoint describes freedom from a DSRC through 6 months and was tested against the null rate of 90%.
Time Frame: 6 months
Population: The Intent-to-Treat Population (ITT) includes all enrolled subjects intended to receive the Cordella PA Sensor who entered the Cath Lab, including those in whom Implant Procedure was not attempted for whatever reason (e.g., Cordella PA Sensor Implant cannot be performed due to anatomical reasons) from the Open Label Arm and Former Treatment Arm. Patients in this population in whom the Cordella PA Sensor Implant was not attempted were followed through 30 days for safety purposes.
Measure: Number (95% Confidence Interval); unit: Proportion of patients without a DSRC
Groups:
- Intent-to-Treat (ITT): Received standard of care heart failure management (i.e., Guideline Directed Medical Therapy) and Pulmonary Artery Pressure Guided Heart Failure Management (PAPGHFM) using the Cordella Heart Failure System (CHFS) with the PA pressure sensor OR withdrew from trial and did not receive an implant.
  Cordella™ Pulmonary Artery Sensor System: The Cordella PA Sensor System (CorPASS) is intended to measure, record, and transmit pulmonary artery pressure (PAP) data from NYHA Class III heart failure patients at home to clinicians for assessment and patient-centered heart failure management and comprises of seven subsystems that operate together to take daily Pulmonary Artery Pressure (PAP) readings at a patient's home and transmit the results to a care provider for evaluation.
  1. Cordella Sensor
  2. Cordella Delivery System
  3. myCordella Patient Reader
  4. Reader Dock
  5. Cordella Calibration Equipment (CalEQ)
  6. myCordella Hub
  7. Cordella Data Analysis Platform (CDAP)
Arm/Group | Intent-to-Treat (ITT) | Former Control Arm
Number analyzed (Participants) | 493 | 72
Proportion of patients without a DSRC | 0.992 [0.979 to 0.997] | 0.986 [0.905 to 0.998]

3. Primary Outcome: Safety: Freedom From Pressure Sensor Failure
Description: A pressure sensor failure (PSF) occurs when the sensor malfunctions to the point that no readings can be obtained from the sensor after all attempts are exhausted including troubleshooting the system to rule out any problems with the electronic components. The second primary safety endpoint describes freedom from Pressure Sensor Failure through 6 months, it was tested against the null rate of 95%.
Time Frame: 6 months
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Proportion of patients without a PSF
Arm/Group | Intent-to-Treat (ITT) | Former Control Arm
Number analyzed (Participants) | 493 | 72
Proportion of patients without a PSF | 0.998 [0.986 to 1.000] | 1.000 [1.000 to 1.000]

4. Secondary Outcome: HF Hospitalizations
Description: Number of HF Hospitalizations at 6 months post-implant compared to the number of HF Hospitalizations in the 6 months prior to implant
Time Frame: 6 Months prior to implant and 6 months post implant
Population: as for outcome 1
Measure: Number; unit: events
Arm/Group | Modified Intent-to-Treat (mITT) | Former Control Arm
Number analyzed (Participants) | 456 | 72
events
  Total HF Hospitalizations events in 6 months before implant | 266 | 36
  Total HF Hospitalizations events in 6 months after implant | 60 | 18
Statistical Analysis 1: Comparison: Modified Intent-to-Treat (mITT); Comparison of HF Hospitalization events 6 months before implant vs 6 months after implant; Test type: Superiority; p < 0.0001, Wilcoxon (Mann-Whitney)

5. Secondary Outcome: HF Hospitalizations or Emergency Department/Hospital Outpatient IV Diuretic Visits.
Description: Incidence rate of HF Hospitalizations, Emergency Department/ Hospital Outpatient IV diuretic visits of Former Control Arm and Modified Intent to Treat at 6 months post implant, added together with equal weighting into a total number of events.
Time Frame: 6 months
Population: The Modified Intent-to-Treat Population (mITT) includes all implanted subjects from the Open Label Armand Former Treatment Arm. All primary and secondary effectiveness analyses are performed on the mITT.
Measure: Number (95% Confidence Interval); unit: Events Per Patient Per 6 Months
Arm/Group | Modified Intent-to-Treat (mITT) | Former Control Arm
Number analyzed (Participants) | 456 | 72
Events Per Patient Per 6 Months | 0.1703 [0.1362 to 0.2130] | 0.2508 [0.1580 to 0.3981]
Statistical Analysis 1: Comparison: Modified Intent-to-Treat (mITT) vs Former Control Arm; Test type: Superiority — Comparison of the incidence rate of HF hospitalizations or emergency department / hospital outpatient IV diuretic visits of Former Control Arm versus Modified Intent to Treat Arm at 6 months post-implant/Subgroup Analysis; p = 0.0697, Poisson Regression

6. Secondary Outcome: Mortality
Description: Cardiac and all-cause mortality
Time Frame: 6 Months
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Modified Intent-to-Treat (mITT) | Former Control Arm
Number analyzed (Participants) | 456 | 72
Participants
  All-cause Mortality | 10 | 2
  Cardiac Mortality | 6 | 2

7. Secondary Outcome: IV Diuretic Visits
Description: Intravenous (IV) diuretic visits
Time Frame: 6 Months
Population: as for outcome 5
Measure: Number; unit: events
Arm/Group | Modified Intent-to-Treat (mITT) | Former Control Arm
Number analyzed (Participants) | 456 | 72
events | 17 | 0

8. Secondary Outcome: Pulmonary Artery Pressure (PAP)
Description: Change in PAP: a. From Baseline through 6 months in subjects with a baseline mPAP i. above target range ii. within or below target range iii. Overall
Time Frame: 6 months
Population: The Modified Intent-to-Treat Population (mITT) includes all implanted subjects from the Open Label Armand Former Treatment Arm. All primary and secondary effectiveness analyses are performed on the mITT. mPAP target was 20 mmHG, thus patients above 20 mmHG for mPAP were assigned to Above Target group and patients at or below 20 mmHG mPAP were assigned to the Within/Below Target group.
Measure: Mean (Standard Deviation); unit: mmHG of mPAP
Groups:
- Modified Intent-to-Treat: The Modified Intent-to-Treat Population (mITT) includes all implanted subjects from the Open Label Armand Former Treatment Arm. All primary and secondary effectiveness analyses are performed on the mITT.
- Above Target mPAP at Baseline: mPAP target was 20 mmHG, thus patients above 20 mmHG for mPAP were assigned to Above Target group.
- Within/BelowTarget mPAP at Baseline: mPAP target was 20 mmHG, thus patients at or below 20 mmHG mPAP were assigned to the Within/Below Target group.
Arm/Group | Modified Intent-to-Treat | Above Target mPAP at Baseline | Within/BelowTarget mPAP at Baseline
Number analyzed (Participants) | 437 | 197 | 240
mmHG of mPAP
  Baseline | 20.2 (10.3) | 29.2 (7.7) | 12.8 (4.9)
  6 Months | 21.4 (9.3) | 26.8 (9.2) | 17.0 (6.8)
Statistical Analysis 1: Comparison: Modified Intent-to-Treat; Test type: Superiority — Comparison of mPAP values at baseline to values at 6 months; p = 0.0952, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Above Target mPAP at Baseline; Test type: Superiority — Comparison of mPAP values at baseline to values at 6 months; p = 0.0090, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Within/BelowTarget mPAP at Baseline; Test type: Superiority — Comparison of mPAP values at baseline to values at 6 months; p < 0.0001, Wilcoxon (Mann-Whitney)

9. Secondary Outcome: Device Success
Description: Proportion of device success as documented by ability of the System to successfully transmit PAP data transmit PAP data
Time Frame: 6 Months
Population: as for outcome 5
Measure: Number; unit: Proportion of device readings successful
Arm/Group | Modified Intent-to-Treat (mITT)
Number analyzed (Participants) | 456
Proportion of device readings successful | 0.991

10. Secondary Outcome: Kansas City Cardiomyopathy Questionnaire (KCCQ)
Description: The Quality of Life KCCQ questionnaire is a measure of health-related quality of life. It is a 23-item, self-administered instrument that quantifies physical function, symptoms (frequency, severity and recent change), social function, self-efficacy and knowledge, and quality of life related to Heart Failure. From 23-items, the Overall Summary Score (OSS) will be calculated. In the OSS, each of the 23 items are converted onto a 0 to 100 scale using this formula: (Raw score - Minimum Raw Score)/(Maximum Raw Score - Minimum Raw Score) * 100. Then these are averaged across the 23 items. A score of 100 (the maximum score) would indicate maximum quality of life relating to heart failure and a score of 0 (scale minimum) would indicate the worst possible quality of life relating to heart failure, with higher scores generally indicating higher quality of life.
Time Frame: 6 Months
Population: All primary and secondary effectiveness analyses are performed on the Modified Intent-to-Treat Population (mITT). For this measure, only patients who completed the measure were included in the results reported, which is the reason for the smaller number of patients in these results than in the mITT population overall.
Measure: Mean (Standard Deviation); unit: points
Arm/Group | Modified Intent-to-Treat (mITT) | Former Control Arm
Number analyzed (Participants) | 421 | 65
points
  Baseline | 52.8 (22.8) | 49.7 (23.8)
  6 Month | 57.8 (24.2) | 54.2 (25.2)
Statistical Analysis 1: Comparison: Modified Intent-to-Treat (mITT); Test type: Superiority — Comparison of KCCQ at baseline and at 6 months; p = 0.0026, Wilcoxon (Mann-Whitney)

11. Secondary Outcome: NYHA
Description: New York Heart Association (NYHA) Classification at 6 months. The New York Heart Association (NYHA) Classification provides a way of classifying the extent of heart failure by classifying patients in one of four categories based on their limitations during physical activity and in degree of shortness of breath and or angina pain. Class I is the least severe and Class IV is the most severe. The classes are:
  Class I - No symptoms and no limitation in ordinary physical activity, e.g. shortness of breath when walking, climbing stairs etc.
  Class II - Mild symptoms (mild shortness of breath and/or angina) and slight limitation during ordinary activity.
  Class III - Marked limitation in activity due to symptoms, even during less-than-ordinary activity, e.g. walking short distances. Comfortable only at rest.
  Class IV - Severe limitations. Experiences symptoms even while at rest. Mostly bedbound patients.
Time Frame: 6 Months
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | Modified Intent-to-Treat (mITT) | Former Control Arm
Number analyzed (Participants) | 414 | 65
Participants
  I | 23 | 3
  II | 121 | 16
  III | 262 | 46
  IV | 8 | 0
Statistical Analysis 1: Comparison: Modified Intent-to-Treat (mITT); The New York Heart Association (NYHA) Classification is a system used to evaluate and classify the severity of heart failure based on symptoms, patient's physical activity, and quality of life. Its scale ranges from class 1 to 4 with class 1 indicating the least severe heart failure symptoms (i.e., the best functionality) and class 4 indicating the most severe heart failure symptoms (i.e., the poorest functionality), with higher classes indicating poorer functioning as relates to heart failure; Test type: Other — Test of difference in distribution of NYHA class from baseline (all patients were class III at baseline); p < 0.0001, Chi-squared

12. Secondary Outcome: 6-Minute Walk Test
Description: Functional status improvement, as measured by 6-Minute Walk Test total distance walked. The 6-Minute Walk Test (6MWT) is a test that measures the total distance an individual can walk on a flat, hard surface in 6 minutes. It is commonly used to evaluate functional exercise capacity in patients with conditions including heart failure. The minimum score possible is 0, which would represent an inability to walk any distance. There is no maximum score, as a patient could theoretically walk any distance in 6 minutes though 800 meters considered the top reference range, which is what would be expected by elite athletes. Higher score indicate greater higher exercise capacity and lower scores indicate lower exercise capacity.
Time Frame: 6 Months
Population: The Modified Intent-to-Treat Population (mITT) includes all implanted subjects from the Open Label Armand Former Treatment Arm. All primary and secondary effectiveness analyses are performed on the mITT. For this measure, only patients who completed the measure were included in the results reported, which is the reason for the smaller number of participants in these results than in the mITT population overall.
Measure: Mean (Standard Deviation); unit: Meters Walked
Arm/Group | Modified Intent-to-Treat (mITT) | Former Control Arm
Number analyzed (Participants) | 436 | 70
Meters Walked
  Baseline | 259.5 (121.1) | 281.5 (133.6)
  6 Months | 283.2 (123.9) | 299.4 (147.5)
Statistical Analysis 1: Comparison: Modified Intent-to-Treat (mITT); Test type: Superiority — Comparison of baseline 6MWT vs 6 month 6MWT; p = 0.1086, Wilcoxon (Mann-Whitney)

13. Secondary Outcome: Number and Percent of Patients With Serious Adverse Events
Description: Number and percent of patients with serious adverse events throughout the study (site-reported).
Time Frame: 6 Months
Population: The Intent-to-Treat Population (ITT) includes all implanted subjects from the Open Label Arm and Former Treatment Arm. All safety analyses were performed on the ITT population.
Measure: Count of Participants; unit: Participants
Arm/Group | Intent-to-Treat (ITT) | Former Control Arm
Number analyzed (Participants) | 493 | 72
Participants
  Subjects with at least one predefined SAE | 196 | 31
  Heart Failure | 79 | 16
  ED Visit | 4 | 0
  Hospitalization | 72 | 16
  Urgent, Unscheduled Outpatient Office/ Practice | 2 | 0
  Acute Kidney Injury (AKIN) | 22 | 7
  Bleeding | 6 | 4
  Conduction Disturbances and Arrhythmias | 28 | 4
  Hemoptysis | 12 | 1
  Myocardial Infarction (MI) | 3 | 1
  Pulmonary Embolism | 6 | 0
  Pulmonary Occlusion | 0 | 0
  Renal Dysfunction | 8 | 1
  Stroke and Trans Ischemic Attach (TIA) | 0 | 1
  Vascular Access Site and Access-Related Complications | 4 | 2
  Vessel Trauma | 4 | 0
  Other | 123 | 17

14. Secondary Outcome: Incidence of HF Hospitalizations or All-cause Mortality
Description: Incidence of HF Hospitalizations or all-cause mortality at 12 months calculated from Poisson regression.
Time Frame: 12 months
Population: Participants who received Cordella PA sensor implant.
Measure: Number (95% Confidence Interval); unit: Events Per Patient Per 12 Months
Arm/Group | Modified Intent-to-Treat (mITT) | Former Control Arm
Number analyzed (Participants) | 456 | 72
Events Per Patient Per 12 Months | 0.3629 [0.3107 to 0.4239] | 0.5438 [0.3957 to 0.7474]

15. Secondary Outcome: N-terminal Pro B-type Natriuretic Peptide (NT-proBNP)
Description: Change of N-terminal pro B-type Natriuretic Peptide (NT-proBNP) from Baseline through 6 months. NT-proBNP is a biomarker used to assess heart failure (HF). NT-proBNP levels vary widely and are reported in picograms per milliliter (pg/mL) or nanograms per liter (ng/L), with no predefined maximum value. Zero is a hypothetical minimum value though this is, in practice, not possible. In the current context, higher scores indicate more severe heart failure and lower levels indicate less severe heart failure.
Time Frame: 6 months
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Modified Intent-to-Treat (mITT) | Former Control Arm
Number analyzed (Participants) | 447 | 70
pg/ml
  Baseline | 1731.4 (3012.8) | 1786.8 (3809.4)
  6 Months | 1632.5 (2742.4) | 1345.6 (2435.7)
Statistical Analysis 1: Comparison: Modified Intent-to-Treat (mITT); Test type: Superiority — Compare NTproBNP at baseline with 6 months; p = 0.0628, Wilcoxon (Mann-Whitney)

16. Secondary Outcome: Days Alive and Out of Hospital (DAOH)
Description: Days Alive and Out of Hospital (DAOH) during the 6 months after implant
Time Frame: 6 Months
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Modified Intent-to-Treat (mITT) | Former Control Arm
Number analyzed (Participants) | 456 | 72
days | 172.0 (27.2) | 173.7 (19.6)

17. Secondary Outcome: Number of Heart Failure Related Medication Changes
Description: Number of patients (%) with heart failure related medication changes in the 6 months after implant
Time Frame: 6 Months
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Modified Intent-to-Treat (mITT) | Former Control Arm
Number analyzed (Participants) | 456 | 72
Participants
  Baseline to 1 Month | 234 | 25
  1 Month to 3 Months | 227 | 25
  3 Months to 6 Months | 260 | 32

18. Secondary Outcome: Number of HF Hospitalization or All-cause Mortality
Description: Number of HF Hospitalizations or all-cause mortality at 12 months
Time Frame: 12 months
Population: Participants who received the Cordella PA sensor implant.
Measure: Number; unit: Events
Arm/Group | Modified Intent-to-Treat (mITT) | Former Control Arm
Number analyzed (Participants) | 456 | 72
Events
  Heart Failure Hospitilizations | 126 | 33
  All-Cause Deaths | 33 | 5

19. Secondary Outcome: Number of HF Hospitalization, Emergency Department/Hospital Outpatient IV Diuretic Visits, All-cause Mortality
Description: Number of combined outcome of:
  1. First and recurrent Heart Failure Hospitalizations
  2. Emergency Department / Hospital Outpatient IV diuretic visits all-cause mortality at 6 months, added together with equal weighting into a total number of events.
Time Frame: 6 months
Population: as for outcome 5
Measure: Number; unit: events
Arm/Group | Modified Intent-to-Treat (mITT) | Former Control Arm | Former Treatment Arm | Open Label Arm
Number analyzed (Participants) | 456 | 72 | 88 | 368
events | 87 | 20 | 17 | 70

20. Secondary Outcome: Number of HF Hospitalization, Emergency Department/Hospital Outpatient IV Diuretic Visits
Description: Number of HF Hospitalization, Emergency Department/Hospital Outpatient IV diuretic visits at 6 months.
Time Frame: 6 months
Population: as for outcome 5
Measure: Number; unit: Events
Arm/Group | Modified Intent-to-Treat (mITT) | Former Control Arm | Former Treatment Arm | Open Label Arm
Number analyzed (Participants) | 456 | 72 | 88 | 268
Events | 77 | 18 | 15 | 62

21. Secondary Outcome: Implant Procedure and Procedure Related Adverse Events and Serious Adverse Events
Description: Frequency of implant procedure and procedure related adverse events and serious adverse events
Time Frame: 6 months
Population: as for outcome 13
Measure: Count of Participants; unit: Participants
Arm/Group | Intent-to-Treat (ITT)
Number analyzed (Participants) | 493
Participants
  Subjects with at least one predefined AE or SAE with study device or implant procedure relationship | 36
  Bleeding | 3
  Conduction Disturbances and Arrhythmias | 4
  Heart Failure | 2
  Hemoptysis | 14
  Pulmonary Embolism | 1
  Vascular Access Site and Access-Related Complications | 12
  Other | 16

ADVERSE EVENTS:
Time Frame: 12 months
Description: The event is an SAE when the patient outcome is:
  * Death
  * Life-threatening
  * Hospitalization (initial or prolonged)
  * Disability or permanent change
  * Congenital Anomaly/Birth Defect
  * Required Intervention to Prevent Permanent Impairment or Damage
  * Other Serious (Important Medical Events) A planned hospitalization for a pre-existing condition, or a procedure required by the protocol, without a serious deterioration in health, is not considered to be a serious adverse event.
Groups:
- Intent-to-Treat (ITT): Received standard of care heart failure management (i.e., Guideline Directed Medical Therapy) and Pulmonary Artery Pressure Guided Heart Failure Management (PAPGHFM) using the Cordella Heart Failure System (CHFS) with the PA pressure sensor OR withdrew from trial and did not receive an implant. To capture safety of all patients in the trial, the ITT sample was used in all safety analyses. In contrast, the mITT sample was used in all efficacy analyses as, as only mITT patients received the active treatment. See participant flow section for more details.
  Cordella™ Pulmonary Artery Sensor System: The Cordella PA Sensor System (CorPASS) is intended to measure, record, and transmit pulmonary artery pressure (PAP) data from NYHA Class III heart failure patients at home to clinicians for assessment and patient-centered heart failure management and comprises of seven subsystems that operate together to take daily Pulmonary Artery Pressure (PAP) readings at a patient's home and transmit the results to a care provider for evaluation.
  1. Cordella Sensor
  2. Cordella Delivery System
  3. myCordella Patient Reader
  4. Reader Dock
  5. Cordella Calibration Equipment (CalEQ)
  6. myCordella Hub
  7. Cordella Data Analysis Platform (CDAP)
Arm/Group | Intent-to-Treat (ITT) | Former Control Arm
All-Cause Mortality (participants affected / at risk) | 33/493 | 5/72
Serious Adverse Events (participants affected / at risk) | 278/493 | 47/72
Other Adverse Events (participants affected / at risk) | 379/493 | 60/72
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intent-to-Treat (ITT) (N=493) | Former Control Arm (N=72)
Heart Failure (Cardiac disorders) | 132 (193) | 23 (58)
Emergency Department Visit (Surgical and medical procedures) | 6 (6) | 0 (0)
Hospitalization (Surgical and medical procedures) | 122 (177) | 23 (58)
Urgent, Unscheduled Outpatient Office/ Practice (Surgical and medical procedures) | 2 (2) | 0 (0)
Acute Kidney Injury (Renal and urinary disorders) | 41 (55) | 8 (11)
Bleeding (Blood and lymphatic system disorders) | 12 (13) | 5 (5)
Conduction Disturbances and Arrhythmias (Cardiac disorders) | 48 (66) | 10 (10)
Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 12 (14) | 1 (1)
Myocardial Infarction (Cardiac disorders) | 6 (6) | 1 (1)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 6 (7) | 1 (1)
Pulmonary Occlusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0)
Renal Dysfunction (Renal and urinary disorders) | 12 (15) | 3 (3)
Stroke and Trans Ischemic Attack (Cardiac disorders) | 2 (2) | 2 (2)
Vascular Access Site and Access-Related Complications (Cardiac disorders) | 4 (4) | 2 (2)
Vessel Trauma (Cardiac disorders) | 4 (4) | 0 (0)
Other (General disorders) | 185 (404) | 24 (61)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intent-to-Treat (ITT) (N=493) | Former Control Arm (N=72)
Blood and lymphatic system disorders (Blood and lymphatic system disorders) | 14 (16) | 6 (7)
Cardiac disorders (Cardiac disorders) | 126 (190) | 18 (29)
Ear and labyrinth disorders (Ear and labyrinth disorders) | 14 (15) | 1 (1)
Gastrointestinal disorders (Gastrointestinal disorders) | 78 (122) | 8 (9)
General disorders and administration site conditions (General disorders) | 83 (113) | 19 (31)
Hepatobiliary disorders (Hepatobiliary disorders) | 7 (7) | 0 (0)
Immune system disorders (Immune system disorders) | 6 (6) | 0 (0)
Infections and infestations (Infections and infestations) | 166 (291) | 28 (45)
Injury, poisoning and procedural complications (Injury, poisoning and procedural complications) | 79 (106) | 14 (25)
Investigations (Investigations) | 49 (60) | 5 (6)
Metabolism and nutrition disorders (Metabolism and nutrition disorders) | 95 (168) | 19 (28)
Musculoskeletal and connective tissue disorders (Musculoskeletal and connective tissue disorders) | 78 (121) | 14 (21)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 12 (15) | 1 (1)
Nervous system disorders (Nervous system disorders) | 72 (111) | 19 (24)
Product issues (Product Issues) | 4 (4) | 0 (0)
Psychiatric disorders (Psychiatric disorders) | 19 (28) | 0 (0)
Renal and urinary disorders (Renal and urinary disorders) | 88 (118) | 18 (29)
Respiratory, thoracic and mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 84 (116) | 14 (20)
Skin and subcutaneous tissue disorders (Skin and subcutaneous tissue disorders) | 28 (32) | 2 (2)
Surgical and medical procedures (Surgical and medical procedures) | 9 (9) | 0 (0)
Vascular disorders (Vascular disorders) | 68 (83) | 12 (16)
Reproductive system and breast disorders (Reproductive system and breast disorders) | 14 (14) | 1 (1)
Endocrine Disorders (Endocrine disorders) | 4 (4) | 0 (0)
Social Circumstances (Social circumstances) | 1 (1) | 0 (0)
Congential, Familial, and Genetic Disorders (Congenital, familial and genetic disorders) | 4 (6) | 0 (0)
Eye Disorders (Eye disorders) | 7 (8) | 1 (1)

LIMITATIONS AND CAVEATS:
* The major limitation of PROACTIVE-HF is its open-label, single arm design and the absence of a concurrent control arm, though endpoint assessment was blinded and performed by an independent adjudication committee
* There are known limitations of interpretation of KCCQ in unblinded studies.
* As prior studies utilized supine PAP for remote management of HF, clinician lack of familiarity with orthostatic PAP physiology may have influenced decision making.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2023-11-08): https://cdn.clinicaltrials.gov/large-docs/59/NCT04089059/Prot_000.pdf
  • Statistical Analysis Plan (2023-08-17): https://cdn.clinicaltrials.gov/large-docs/59/NCT04089059/SAP_001.pdf